CLINICAL TRIAL: NCT03132051
Title: Sonographic Evaluation of Patients With Carpal Tunnel Syndrome Following Steroid Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-07-006A; 2012-05-021A
Record Dates: First submitted 2017-02-16; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Steroids; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: All patients received steroid injection for carpel tunnel syndrome (CTS) and ultrasonographic evaluation before and after steroid injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- steroid injection (Experimental): ultrasound-guided steroid injection using 1ml of 10 mg (10mg/ml) triamcinolone acetonide
  Interventions: Drug: steroid injection

INTERVENTIONS:
Drug: steroid injection — ultrasound-guided steroid injection using 1ml of 10 mg (10mg/ml) triamcinolone acetonide
  Other Names: triamcinolone acetonide

SUMMARY:
The objective of this study was to assess sonographic changes of the median nerve after steroid injection for carpal tunnel syndrome.

DETAILED DESCRIPTION:
Patients with CTS were recruited. The Boston Questionnaire (BQ) was administered and ultrasonographic and electrophysiological examinations were performed before and at two, six, and 12 weeks after steroid injection. Cross sectional area (CSA) was measured at 2 levels: at the tunnel inlet and in the mid-carpal tunnel. Flattening ratio (FR) was measured only in the mid-carpal tunnel. Correlation analyses between baseline ultrasonography, BQ, and electrophysiological measures were performed.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of CTS
2. The diagnosis of CTS was confirmed by electrophysiological tests.

Exclusion Criteria:

1. neurologic disorders that could mimic CTS such as cervical radiculopathy, polyneuropathy, proximal median nerve entrapment, or thoracic outlet syndrome
2. history of distal radius fracture
3. pregnancy or lactation
4. regular use of systemic NSAIDs or corticosteroids
5. known allergy to corticosteroids and local anesthetics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Cross sectional area | 12 weeks
  The CSA of the median nerve was measured at 2 levels: at the carpal tunnel inlet (CSA-I; immediately prior to the proximal margin of the flexor retinaculum) and in the mid-carpal tunnel (CSA-M; at the level of the pisiform bone and scaphoid tubercle)

SECONDARY OUTCOMES:
flattening ratio | 2, 6, 12 weeks
  The flattening ratio was measured only at the mid-tunnel (FR-M). FR was calculated by dividing the horizontal diameter of the nerve by the vertical diameter.
Boston Carpal Tunnel Questionnaire (BQ) | 2, 6, 12 weeks
  The BQ was interviewed-administered to assess the severity of symptoms and functional status.
Median nerve distal motor latency | 2, 6, 12 weeks
  the CMAPs were obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode was placed on the muscle belly, and the reference electrode was placed on the tendon insertion. The median nerve was stimulated 8 cm proximal to the active recording electrode. Distal motor latencies were measured from the onset of stimulus artifact to the onset of the CMAP
sensory nerve conduction velocity | 2, 6, 12 weeks
  SNAPs were obtained using an antidromic method and recorded by surface electrodes placed at the proximal and distal interphalangeal joints of the index finger for the median nerve and the same joints of the little finger for the ulnar nerve. The median nerves were stimulated at the wrist at a distance of 14 cm from the wrist to the active electrode. Distal sensory latencies were measured from the onset of the stimulus artifact to the onset of the SNAP. SNCV was calculated dividing the distance of 14 cm by the distal sensory latency.
compound muscle action potential amplitude (CMAP) | 2, 6, 12 weeks
  the CMAPs were obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode was placed on the muscle belly, and the reference electrode was placed on the tendon insertion. The median nerve was stimulated 8 cm proximal to the active recording electrode. The amplitude of CMAP were measured from baseline to negative peak.
sensory nerve action potential amplitudes. | 2, 6, 12 weeks
  SNAPs were obtained using an antidromic method and recorded by surface electrodes placed at the proximal and distal interphalangeal joints of the index finger for the median nerve and the same joints of the little finger for the ulnar nerve. The median nerves were stimulated at the wrist at a distance of 14 cm from the wrist to the active electrode. The amplitude of SNAP were measured from baseline to negative peak.

CONTACTS AND LOCATIONS:
Overall Officials: Jia chi Wang, Principal Investigator — Taipei Veteran General hospital
Locations (1):
- Teipei Veterans General Hospital, Taipei, Taiwan